CLINICAL TRIAL: NCT01192607
Title: Endoscopic Treatment During Endodontic Procedures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: oded nahlieli, OMFS BARZILAI MEDICAL CENTER
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTA3741; BAR1404CTIL
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2011-03

CONDITIONS: Dental Pulp Cavity; Root Canal Treatment; Endoscopy
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endoscopic treatment during root canal treatment — Endoscopic treatment during root canal treatment

SUMMARY:
The objectives of this Phase I study is to evaluate the safety and effectiveness of the endoscopic endodontic equipment device for root canal assistance treatment as well as to evaluate the ease of use of this device, by a surgeon experienced in endodontic treatment, in a true clinical setting.

DETAILED DESCRIPTION:
This open, phase 1 trial will be conducted on 15 patients with the need for root canal treatment. The teeth will be permanent teeth in which the need for root canal treatment was decided by his dentist in the dental clinic in the Barzilai medical center Ashkelon. Videoendoscopy of the procedure will be recorded and will include a post-op view of the treatment. Patients will be followed up for pain infection and any potential complications; immediately, at 4 weeks 12 weeks and 6 month post- op. The procedure will also be taped externally to document surgeon's convenience with the equipment.

The procedures will be performed under local or general anesthesia in an ambulatory environment, using standard root canal equipment, which will include endodontic hand and rotary files, endodonically used irrigating solutions and the videoendoscopy equipment. Under this protocol the basic treatment will be carried out by professional well trained endodontist in the same way used for root canal treatment. Following the mechanical preparation of the canal the endoscope, connected to a video camera and monitor, is introduced with the help of isotonic saline irrigation. With the aid of the endoscope remains of soft tissue from the pulp tissue will be coagulated with the ERBOTOM ICC 80 monopolar fibers and removed with the irrigation, the canal will be inspected for lateral canals and the monoplar fibers will be used for coagulating and removal of this tissue. Er-Yag laser fiber connected to Erbium laser generator will be used for finalizing the canal preparation and preparation of the lateral canals. Actual lasing and coagulation will be performed only under clear vision, when the fiber is seen to be in direct contact with the tissue. Adequate irrigation will be maintained throughout the procedure using an intravenous bag connected to the irrigation port on the sheath of the endoscope.

The endoscope device will be connected to the Erbbe diathermy ERBOTOM ICC 80 for coagulation monopolar fibers 0.05-0.1 mm number 20197-021-022 .

Standard Lumenis Opus 20, dental Erbium:YAG laser available in the hospital. Lasing will begin at a setting of 300 mj per pulse and a pulse rate of 7 Hz.

The same procedures performed on 15 human teeth in a lab status. The insertion of the instruments to the root canal will be in 2 techniques:1) Via the endoscope channel and 2) The instruments will be inserted parallel to the endoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. Suffers from deep carries, acute or chronic pulpitis crown fracture which root canal treatment is the treatment of choice.
3. Patient understands and has signed the Informed Consent Form.

Exclusion Criteria:

1. Teeth with cracks or root fracture.
2. Patients on anti-coagulants.
3. Patients with cardiac diseases, kidney insufficiency, any malignancy or any steroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Endoscopic root canal treatment | 1 month

SECONDARY OUTCOMES:
Endoscopic root canal complications | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Oded Nahlieli, DMD, Principal Investigator — Barzilai Medical Center
Locations (1):
- Oral and Maxillofacial Surgery, Barzilai Medical Center, Ashkelon, Israel